CLINICAL TRIAL: NCT06047847
Title: Determination of Biological Activity of Enriched Serum Among Healthy Participants After Consumption of the Food Supplement TOTUM-448
Brief Title: Determination of Biological Activity of Enriched Serum Following TOTUM-448 Consumption
Acronym: CnC-TOTUM448
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: Clinic'n'Cell (Other); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-A00579-36
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: NAFLD; MASLD; Mild Inflammatory Context
Keywords: ex vivo; lipid metabolism; inflammation; hepatocytes; oxidative stress; plant extract; polyphenols; dietary/food supplement
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Inflammation

STUDY DESIGN:
Intervention Model Description: An ex vivo clinical approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOTUM-448 (Experimental): 10 healthy men will consume an acute intake of 4.284g of TOTUM-448 on three separate occasions.
  Phase 1: once per galenic form (capsule and powder). Phase 2: once (capsule only).
  Interventions: Dietary Supplement: TOTUM-448

INTERVENTIONS:
Dietary Supplement: TOTUM-448 — The study is divided in two phases. The first clinical phase of the project is aimed at determining TOTUM-448's metabolites absorption peak (two galenic forms will be tested: capsules and powder). Then, human circulating metabolites from polyphenols will be quantified and characterized by ultra-high performance liquid chromatography hyphenated with tandem mass spectrometry (UPLC-MS/MS). Once the absorption profile is characterized, volunteers will visit once again the clinical center for the collection of serum fractions either naïve (before ingestion) or enriched (containing circulating metabolites following TOTUM-448 ingestion). The enriched fraction (circulating bioactive collection) will be collected at t-max as characterized in the first phase (absorption profil's peak). Finally, biological activity of TOTUM-448 on human hepatocytes will be studied by comparing naïve serum and serum containing circulating metabolites according to an in vitro protocol.

SUMMARY:
Dietary intakes of saturated fatty acids remain well above nutritional recommendations for most European countries. This may progressively lead to a pro-inflammatory context and the alteration of lipid metabolism in the liver. The hypothesis of this study is that TOTUM-448 promotes the normal function of hepatocytes in a mild inflammatory context. To determine the cellular and molecular effects of TOTUM-448, circulating bioactive molecules after TOTUM-448 intake will be collected and then studied in human hepatocytes using an innovative ex vivo clinical approach developed by Clinic'n'Cell.

ELIGIBILITY:
Main Inclusion Criteria:

* Lipid profile within reference values
* Glycemia < 100mg/dL
* Normal hepatic function
* Normal blood formulation
* Normal renal function
* BMI between 20 and 28kg/m2
* Non smoker or occasional smoker

Main Exclusion Criteria:

* All types of vaccination within one month
* Alcohol intakes superior to World Health Organization recommendations
* Ongoing pharmacological, dietary supplement and/or probiotic treatment
* Consumption of enriched functional foods or dietary supplements within two weeks of inclusion
* Any known disease
* Allergy to ingredients of the study product
* With dietary habits incompatible with the study conduct

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the influence of circulating bioactive metabolites in blood stream resulting from the intake of TOTUM-448 on viability of human hepatocytes in a hyperlipidic pro-inflammatory context. | At phenolic compounds t-max obtained during kinetic phase. Note: According to previous studies, t-max is expected around 60 minutes.
  Naïve will be compared to enriched serum from the 10 healthy participants at the previously determined t-max.
Evaluate the influence of circulating bioactive metabolites in blood stream resulting from the intake of TOTUM-448 on cholesterol storage of human hepatocytes in a hyperlipidic pro-inflammatory context. | At phenolic compounds t-max obtained during kinetic phase. Note: According to previous studies, t-max is expected around 60 minutes.
  Naïve will be compared to enriched serum from the 10 healthy participants at the previously determined t-max.
Evaluate the influence of circulating bioactive metabolites in blood stream resulting from the intake of TOTUM-448 on triglyceride storage of human hepatocytes in a hyperlipidic pro-inflammatory context. | At phenolic compounds t-max obtained during kinetic phase. Note: According to previous studies, t-max is expected around 60 minutes.
  Naïve will be compared to enriched serum from the 10 healthy participants at the previously determined t-max.
Evaluate the influence of circulating bioactive metabolites in blood stream resulting from the intake of TOTUM-448 on oxidative stress status of human hepatocytes in a hyperlipidic pro-inflammatory context. | At phenolic compounds t-max obtained during kinetic phase. Note: According to previous studies, t-max is expected around 60 minutes.
  Naïve will be compared to enriched serum from the 10 healthy participants at the previously determined t-max.
Evaluate the influence of circulating bioactive metabolites in blood stream resulting from the intake of TOTUM-448 on pro-inflammatory cytokine expression of human hepatocytes in a hyperlipidic pro-inflammatory context. | At phenolic compounds t-max obtained during kinetic phase. Note: According to previous studies, t-max is expected around 60 minutes.
  Naïve will be compared to enriched serum from the 10 healthy participants at the previously determined t-max.

SECONDARY OUTCOMES:
Time to reach the maximum concentration in serum of detectable polyphenol metabolite concentrations by UPLC-MS/MS. | From timepoint 0 minute to timepoint 240 minutes.
  After ingestion of TOTUM-448 the concentration in serum of detectable polyphenol metabolites will be assessed every 20 minutes during 240 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- University Hospital Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wauquier F, Boutin-Wittrant L, Krisa S, Valls J, Langhi C, Otero YF, Sirvent P, Peltier S, Bargetto M, Cazaubiel M, Sapone V, Bouchard-Mercier A, Roux V, Macian N, Pickering G, Wittrant Y. Circulating Human Metabolites Resulting from TOTUM-070 Absorption (a Plant-Based, Polyphenol-Rich Ingredient) Improve Lipid Metabolism in Human Hepatocytes: Lessons from an Original Ex Vivo Clinical Trial. Nutrients. 2023 Apr 14;15(8):1903. doi: 10.3390/nu15081903. PMID 37111121